CLINICAL TRIAL: NCT05093231
Title: A Phase II Study Combining Pembrolizumab With Olaparib in Metastatic Pancreatic Adenocarcinoma (PDA) Patients With Mismatch Repair Deficiency or Tumour Mutation Burden > 4 Mutations/Mb
Brief Title: Pembrolizumab With Olaparib as Combined Therapy in Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Pippa G Corrie, PhD FRCP, Chief Investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PemOla
Record Dates: First submitted 2021-06-03; First posted 2021-10-26 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
Keywords: High tumour burden; molecular profiling; confirmed MMRD or MSI-H IHC; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab and olaparib (Experimental): Pembrolizumab will be given as a fixed dose of 200mg standard dose on Day 1 (+/-3 days) of every 3 weeks cycle , administered intravenously as a ~30 minute infusion, as per standard clinical practice.
  Olaparib dose is 300mg given orally, twice daily, from Day 1 to Day 21 continuously of each 3-week cycle. Dosing will start on day 1 of each cycle.
  Interventions: Drug: Pembrolizumab; Drug: Olaparib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is a highly selective immunoglobulin G4-kappa humanised monoclonal antibody against Programmed cell death protein 1 (PD-1) receptor. It was generated by grafting the variable sequences of a very high-affinity mouse antihuman PD-1 antibody onto a human IgG4-kappa isotype with the containing a stabilizing Serine 228 to Proline Fc mutation.
  Other Names: Keytruda; MK-3475
Drug: Olaparib — Olaparib is a potent inhibitor of polyadenosine 5'diphosphoribose polymerase (PARP) developed as a monotherapy as well as for combination with chemotherapy, ionising radiation and other anti-cancer agents including novel agents and immunotherapy.
  Other Names: Lynparza; AZD2281; KU-0059436

SUMMARY:
A phase II study combining pembrolizumab with olaparib in metastatic pancreatic adenocarcinoma patients with high tumour mutation burden

DETAILED DESCRIPTION:
This is a phase II single arm, open label, prospective trial investigating the efficacy of pembrolizumab plus olaparib in metastatic pancreatic adenocarcinoma patients exhibiting high tumour mutation burden (defined as ≥4 mutations/Mb, including tumours with Mismatch Repair Deficient (MMRD) /Microsatellite Instability (MSI) high).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Written informed consent
* Histologically or cytologically confirmed PDA
* Confirmation that the PDA has TMB >4 mutations/Mb, or dMMR gene mutation, or MSI-H by IHC. TMB status and dMMR can be obtained from either tissue, or blood.
* Radiologically confirmed stage 4 mPDA, with measurable disease
* Received no more than 1 prior systemic therapy regimen for unresectable (stage 3 or 4) PDA is allowed
* Measurable disease which has not been irradiated in prior radiotherapy
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* Life expectancy >12 weeks from the date of screening assessment
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) ≥1.5 x 109 /L
  * Haemoglobin (Hb) ≥ 90 g/L
  * Platelets ≥100 x 109 /L
* Adequate liver function:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤2.5 x upper limit of normal range (ULN), or <5 x ULN in the presence of liver metastases
  * Total bilirubin <1.5 x ULN
* Adequate renal function defined as a calculated creatinine clearance by Cockcroft - Gault of ≥50 mL/min

Exclusion Criteria:

* Patients with resectable or locally advanced PDA
* Other invasive malignancies diagnosed within the last 2 years which have not been treated with curative intent
* Prior immune checkpoint inhibitors or PARP inhibitors. This includes any prior therapy with an anti-PD-1, or anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g, CTLA-4, OX 40, CD137)
* Requirement for non-physiological dose of daily oral steroids, or regular use of any other immunosuppressive agents; prednisolone dose of < 10mg (or equivalent steroid dose) is allowed. Use of inhaled or topical steroids is allowed.
* Significant acute or chronic medical or psychiatric condition, disease or laboratory abnormality, which in the judgment of the investigator would place the patient at undue risk or interfere with the trial. Examples include, but are not limited to:

  * A history of chronic obstructive pulmonary disease, interstitial lung disease, sarcoidosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, cystic fibrosis or bronchiectasis affecting pulmonary function, causing breathlessness at rest
  * Uncontrolled ischaemic heart or other cardiovascular event (myocardial infarction, new angina, stroke transient ischaemic attack, or new congestive cardiac failure) within the last 2 months
  * Stable but significant cardiovascular disease defined by heart failure (New York Heart Association Functional Classification III or IV) or frequent angina
  * Presence of active infection
  * Cirrhotic liver disease, known HIV, chronic active or acute hepatitis B, or hepatitis C
  * History of severe allergy or hypersensitivity reactions
  * Autoimmune disease requiring chronic use of immunosuppressive agents.
  * Replacement therapy using physiological doses for adrenal or pituitary insufficiency is allowed.
  * Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
  * Has known brain metastases and/or carcinomatous meningitis
  * Has myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML.
* Women who are pregnant, or plan to become pregnant or are lactating.
* Women of child-bearing potential and male patients who are unwilling to adhere to the contraception requirement from informed consent until the last dose of the trial treatment and for 120 days after the last dose of trial treatment.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the trial medication.
* Concomitant use of known potent CYP3A4 inhibitors and inducers. Restrictions relating to concomitant medications are described in section 10.9. Please consider wash-out periods.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to screening.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
* Participant received colony-stimulating factors (e.g., granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM CSF] or recombinant erythropoietin) within 28 days prior to the first dose of study intervention.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Participant has persistent toxicities (>CTCAE Grade 2) caused by previous cancer therapy, excluding alopecia.
* Has had an allogenic tissue/solid organ transplant
* Judgment by the Investigator that the patient should not participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, an average of 2 years
  ORR assessed by (RECIST) version 1.1 and CT scanning every 9 weeks for the first 9 cycles (27 weeks), then 12 weekly

SECONDARY OUTCOMES:
Incidence of adverse events (Safety and toxicity) | Through study completion, an average of 2 years
  Safety and toxicity using NCI CTCAE version 5.0
Duration of Response (DOR) | Through study completion, an average of 2 years
  DOR: the time (in days) from the first documentation of objective response (complete response or partial response, confirmed or unconfirmed, whichever status was recorded first, using RECIST criteria) until the first documented disease progression, or death (if before progression
Progression Free Survival (PSF) | through study completion, a maximum of 2 years
  PFS: the time from registration to disease progression, or death, whichever occurs first, assessed by the treating investigators. Patients who remained alive without disease progression at the time of data analyses are censored at their last date of clinical follow-up for progression. Median, 1 year and 2 year PFS rates will be measured
Overall survival (OS) | through study completion, a maximum of 2 year
  OS: the time from registration to death. Patients who remain alive are censored at their last contact date for OS. Median, 1 year and 2 year OS rates will be measured.
European Organisation for Research and Treatment of Cancer Quality of Life of Cancer Patients questionnaire (EORTC QLQC30) | Every 9 weeks during the first 27 weeks and then every 12 weeks until death or maximum of 2 years
  EORTC QLQC30 quality of life questionnaire. Min score 28, maximum score 112. Higher scores equal worse outcome. (Extra 2 questions: min score 1, max score 7 each. Higher scores equals better outcomes.)
European Organisation for Research and Treatment of Cancer Pancreatic Cancer Quality of Life Questionnaire (EORTC PAN26) | Every 9 weeks during the first 27 weeks and then every 12 weeks until death or maximum of 2 years
  EORTC PAN26 quality of life questionnaire. Min score 26, maximum score 104. Higher scores equals worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Corrie, Principal Investigator — Cambridge University Hospital
Locations (13):
- United Kingdom (13):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Velindre Cancer Centre, Cardiff
  - University Hospitals Coventry and Warwickshire, Coventry
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James' University Hospital, Leeds
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Free Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie, Manchester
  - Milton Keynes University Hospital, Milton Keynes
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham University Hospitals NHS Foundation Trust, Nottingham
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No